CLINICAL TRIAL: NCT04144439
Title: Effect of Gamma Aminobutyric Acid on ADHD and Seizures in Children With Epilepsy.
Brief Title: Effect of GABA on ADHD and Seizures in Children With Epilepsy.
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Sherief Abd-Elsalam (Other)
Responsible Party: Sponsor-Investigator, Sherief Abd-Elsalam, Ass. Prof. Tropical Medicine, Tanta University
Organization: Tanta University (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GABA
Record Dates: First submitted 2019-10-04; First posted 2019-10-30 (Actual); Last update posted 2019-10-30 (Actual); Status verified 2019-10

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — gamma-Aminobutyric Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Before treatment (No Intervention): no intervention
- After treatment (Active Comparator): GABA
  Interventions: Drug: GABA

INTERVENTIONS:
Drug: GABA — Gamma amino butyric acid
  Other Names: Gamma amino butyric acid
  Arms: After treatment

SUMMARY:
Effect of GABA on ADHD and seizures in Children with epilepsy.

DETAILED DESCRIPTION:
Effect of Gamma aminobutyric acid on ADHD and seizures in Children with epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* Epilepsy
* ADHD

Exclusion Criteria:

* Epilepsy without ADHD

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2028-12-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Number of seizures | 6 months
  Number of seizures

CONTACTS AND LOCATIONS:
Overall Officials: Abeer Salamah, Lecturer, Principal Investigator — Lecturer of Pediatrics - Kafr Elsheikh University
Locations (1):
- Sherief Abd-Elsalam, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No